CLINICAL TRIAL: NCT02220712
Title: A Multicenter Open-label Study Investigating the Pharmacokinetics and Safety of Aripiprazole IM Depot Formulation (OPC-14597 IMD) During Repeated Administration by Injection Into the Deltoid Muscle in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 031-13-005; JapicCTI-142635 (Other: Japic)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; Deltoid
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: OPC-14597 IMD (Experimental)
  Interventions: Drug: OPC-14597 IMD

INTERVENTIONS:
Drug: OPC-14597 IMD — Administration by injection into the deltoid muscle for a total of 5 doses of 400 mg in 4-week intervals

SUMMARY:
To assess the pharmacokinetics and safety of aripiprazole intra-muscular (IM) depot formulation in patients with schizophrenia after repeated administration by injection into the deltoid muscle for a total of 5 doses of 400 mg in 4-week intervals

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual (DSM)-IV-Text Revision (TR) (295.30, 295.10, 295.20, 295.90, 295.60)
* Patients who have provided written informed consent by themselves (If the patient is a minor, written consent from a legal representative must be obtained in addition to the patient's own written informed consent.)
* Patients, both male and female, aged 18 years or older, but younger than 65 years, at the time of obtaining informed consent
* Patients with a body mass index of 18.5 or higher and lower than 35.0
* Patients whose mental condition is stable or well maintained for 2 weeks or more without any change to dosage regimen for their non-aripiprazole oral atypical antipsychotic monotherapy prior to obtaining informed consent
* Patients who have received aripiprazole in the past

Exclusion Criteria:

* Patients diagnosed as having a mental disorder other than schizophrenia, as defined by DSM-IV-TR criteria.
* Patients with a history or complication of diabetes.
* Patients with hepatic, renal, cardiac, or hematopoietic disorders.
* Female patients who are pregnant or lactating, who may possibly be pregnant, who wish to become pregnant, or male patients whose partner wishes to become pregnant.
* Patients who have a drug allergy or drug hypersensitivity
* Patients for whom clozapine has been ineffective, patients who have responded only to clozapine, or patients who are currently being treated with clozapine.
* Patients with a complication of Parkinson's Disease (excluding drug-induced Parkinsonism).
* Patients with a history or a complication of neuroleptic malignant syndrome, rhabdomyolysis, tardive dyskinesia, paralytic ileus or water intoxication.
* Patients with a history or a complication of psychological or behavioral abnormalities associated with use of psychoactive substances (abuse of alcohol, narcotics, or organic solvent, etc).
* Patients with a history or a complication of suicide attempt or self-injury within 52 weeks prior to obtaining informed consent.
* Patients with a history of or a complication of convulsive disorder such as epilepsy.
* Patients with a history of or a complication of organic brain disorder including cerebrovascular disease.
* Patients with a history or a complication of granulocytopenia or agranulocytosis.
* Patients who have received electro-convulsive therapy (ECT) within 12 weeks prior to obtaining informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPC-14597 IMD
Started | 17
Completed | 13
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Exacerbation of symptoms of an underlying disease | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included subjects who received aripiprazole IMD at least once and who had safety data after aripiprazole IMD administrationn.
Arm/Group | OPC-14597 IMD
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 17
Region of Enrollment [Number; unit: participants]
  Japan | 17

OUTCOME MEASURES:

1. Primary Outcome: OPC-14597 Plasma Concentration 672 Hours Postdose Following Multiple Administration of OPC-14597 IMD Injections
Time Frame: 672 hours postdose of the first, second, third, fourth, and fifth IMD injections
Population: Pharmacokinetic analysis set included subjects whose plasma concentrations were measured without deviation at all blood sampling timepoints during the OPC-14597 IMD treatment period.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- OPC-14597 IMD (First Dose); OPC-14597 IMD (Second Dose); OPC-14597 IMD (Third Dose); OPC-14597 IMD (Fourth Dose); OPC-14597 IMD (Fifth: Administration by injection into the deltoid muscle for a total of 5 doses of 400 mg in 4-week intervals
Arm/Group | OPC-14597 IMD (First Dose) | OPC-14597 IMD (Second Dose) | OPC-14597 IMD (Third Dose) | OPC-14597 IMD (Fourth Dose) | OPC-14597 IMD (Fifth
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
ng/mL | 91.9 (29.4) | 141 (54.0) | 171 (76.1) | 198 (102) | 201 (88.9)

ADVERSE EVENTS:
Time Frame: 20 weeks of treatment period + posttreatment observation period (57 days after administration of the fifth IMD)
Description: Only treatment-emergent adverse events (TEAEs) were assessed for this trial.
Arm/Group | OPC-14597 IMD
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-14597 IMD (N=17)
Schizophrenia (Psychiatric disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-14597 IMD (N=17)
Nasopharyngitis (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Headache (Nervous system disorders) | 2
Dyskinesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Injection site pain (General disorders) | 6
Injection site induration (Gastrointestinal disorders) | 2
Injection site swelling (General disorders) | 2
Injection site erythema (General disorders) | 1
Injection site discomfort (General disorders) | 1
Weight increased (Investigations) | 3
Blood glucose increased (Investigations) | 1
Blood insulin increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No